CLINICAL TRIAL: NCT02546557
Title: Assessment of the Performance of a New Suture Material (Optilene® Suture) for Coronary Artery Bypass Graft Surgery. An Observational Post CE-mark Study
Brief Title: Optilene® Suture for Coronary Artery Bypass Graft Surgery
Acronym: OPTICABG
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1421
Record Dates: First submitted 2015-08-11; First posted 2015-09-11 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Coronary Heart Disease; Multi Vessel Coronary Artery Disease
Keywords: CABG; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Coronary Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OPTICABG: Patients undergoing a coronary artery bypass graft surgery for the repair of a multi-vessel disease or left main-coronary disease.
  Interventions: Procedure: Coronary Artery Bypass Graft surgery

INTERVENTIONS:
Procedure: Coronary Artery Bypass Graft surgery

SUMMARY:
The study is a voluntary study, initiated by B. Braun to collect clinical data for Optilene® suture concerning its key indication.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery is one of the most common elective surgical procedure. In total 40.000 CABG´s have been performed yearly in Germany in 2012 and 2013 which presents 60% of all cardiac surgical interventions. Coronary artery bypass grafting is performed for patients with coronary artery disease (CAD) to improve quality of life and to reduce cardiac-related mortality. CAD is the most leading cause of mortality in the Western world as well as in developing countries and it is the most common cause of heart failure. CABG was introduced in the 1960s. CABG operation has become the most studied intervention in the history of surgery. It is highly effective in the treatment of severe angina and it delays unfavorable events such as death, myocardial infarction and recurrence of angina in comparison to other treatment forms. There is a general agreement that already in the early postoperative period CABG surgery improves the disease in patients with symptomatic left main coronary artery stenosis or stenosis of the three main coronary vessels.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective primary coronary artery bypass graft surgery (CABG).
* On pump or off pump CABG surgery
* Age ≥25 years
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Insulin dependent Diabetes Mellitus
* Acute myocardial infarction with Creatinine Kinase-MB level > 10% of CK and /or ECG signs
* Known immunodeficiency or immunosuppression
* Other combined aortic valve intervention except cardiac valve or mitral valve surgery
* Participation or planned participation in another cardiovascular study before study follow-up is completed.
* Inability to give informed consent due to mental condition, mental retardation, or language barrier.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
postoperative CABG adverse events in hospital | day of discharge (average 7 to 10 days)
  Incidence of individual postoperative CABG adverse events in hospital. Postoperative CABG adverse events are defined as the sum of the frequency of myocardial infarction, stroke, mortality, renal failure and gastrointestinal bleeding.

SECONDARY OUTCOMES:
Incidence of myocardial infarction (MI) | until day of discharge (average 7 to 10 days), 30 days and 3 months postop
Incidence of stroke | until day of discharge (average 7 to 10 days), 30 days and 3 months postop
Mortality | until day of discharge (average 7 to 10 days), 30 days and 3 months postop
Gastrointestinal bleeding | until day of discharge (average 7 to 10 days)
Incidence of renal failure | until day of discharge (average 7 to 10 days)
Anastomosis revision rate due to rebleeding | until day of discharge (average 7 to 10 days)
Other adverse events (wound infection, angina, reoperation) | until 3 months postop

OTHER OUTCOMES:
Repeat Revascularization | until 1 and 3 months postop
  Incidence of repeat revascularization leading to CABG or Percutaneous Coronary Intervention (PCI)
Handling of the suture material | at time of surgery
  Handling of the suture material using a questionnaire containing different dimension and a 5 point assessment level (Likert Scale)
Length of the postoperative hospital stay | Until discharge (average 7 to 10 days)
Improvement of Quality of life Score (EQ-5D-5L) | 3 months postop

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Padró, Prof. Dr., Principal Investigator — Hospitla de la Santa Creu I Sant Pau
Locations (4):
- Robert Bosch KH Stuttgart, Stuttgart, Germany
- Sacco Hospital, Milan, Italy
- Hospital de Santa Maria, Lisbon, Portugal
- Hospital de la Santa Creu I Sant Pau, Barcelona, Spain

REFERENCES:
- [Background] Hawkes AL, Nowak M, Bidstrup B, Speare R. Outcomes of coronary artery bypass graft surgery. Vasc Health Risk Manag. 2006;2(4):477-84. doi: 10.2147/vhrm.2006.2.4.477. PMID 17323602
- [Result] Ursulescu A, Baumann P, Ferrer MT, Contino M, Romagnoni C, Antona C, Padro Fernandez JM. Optilene, a new non-absorbable monofilament is safe and effective for CABG anastomosis. OPTICABG - A prospective international, multi-centric, cohort study. Ann Med Surg (Lond). 2018 Sep 15;35:13-19. doi: 10.1016/j.amsu.2018.09.005. eCollection 2018 Nov. PMID 30258627